CLINICAL TRIAL: NCT06019403
Title: Association Between a Healthy Lifestyle Behavior and Musculoskeletal Pain: an Online Cross-sectional Survey
Brief Title: Association Between a Healthy Lifestyle Behavior and Musculoskeletal Pain
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Other Study IDs: MUSKULO PAIN
Record Dates: First submitted 2023-08-16; First posted 2023-08-31 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Neck Pain; Low Back Pain; Temporomandibular Pain
Keywords: Lifestyle; Cross-sectional; Musculoskeletal pain; Survey
MeSH Terms: conditions — Neck Pain; Low Back Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People without musculoskeletal pain: People who do not suffer from musculoskeletal pain (neck pain, low back pain and/or temporomandibular pain), with or without a healthy lifestyle behavior.
- People with musculoskeletal pain: People suffering from musculoskeletal pain (neck pain, low back pain and/or temporomandibular pain), with or without a healthy lifestyle behavior.

SUMMARY:
Objective: The aim of this online cross-sectional survey is to determine the association between a combination of lifestyle factors and the presence of musculoskeletal pain (neck pain, low back pain and/or temporomandibular pain), in the Belgian adult population.

Methods: Belgian adults from the general population will be recruited using non-probability sampling (convenience and snowballing). The survey will be available online for a period of 6 months on LimeSurvey software. Multivariable logistic regression analyses will be performed to determine the association between a combination of lifestyle factors (sleep, physical activity, stress, weight, smoking, nutrition) and the presence of musculoskeletal pain.

Discussion: The results of the study will provide data about associations between a combination of lifestyle factors and the presence of musculoskeletal pain. This could strengthen current evidence about the importance of adhering to a healthy lifestyle and improve understanding of its association with musculoskeletal pain.

DETAILED DESCRIPTION:
Background: Numerous studies have evaluated the association between some lifestyle factors (e.g., physical activity, sleep, stress) and the presence of musculoskeletal pain (neck pain, low back pain or temporomandibular pain). However, the vast majority of them studied only one lifestyle factor at a time, included specific populations (e.g., workers, nurses), or did not use validated questionnaires. Very few studies to date have investigated the combination of several lifestyle factors. Assessing a single factor does not represent reality, since lifestyle factors are correlated with each other (adherence to some encourages adherence to others, as does non-adherence).

Objective: The aim of this online cross-sectional survey is to determine the association between a combination of lifestyle factors and the presence of musculoskeletal pain (neck pain, low back pain and/or temporomandibular pain), in the Belgian adult population.

Methods: Belgian adults from the general population will be recruited using non-probability sampling (convenience and snowballing). The survey will be available online for a period of 6 months on LimeSurvey software. The questionnaire will include questions about general data, presence of musculoskeletal pain (neck pain, low back pain and temporomandibular pain), and lifestyle factors (sleep, physical activity, stress, weight, smoking, nutrition). Multivariable logistic regression analyses will be performed to determine the association between the combination of lifestyle factors and the presence of musculoskeletal pain. Musculoskeletal pains (neck, low back, temporomandibular) will be analyzed separately and together (multisite pain). As sex seems to play a role in the presence of musculoskeletal pain, different analyses will be performed according to sex (both sexes, males only, females only). Potential confounding and modifying factors (e.g., age, anxiety, depression,...) will be included in the multivariable logistic regression models. Results will be presented using odds ratios (OR) and their 95% confidence intervals.

Discussion: The results of the study will provide data about associations between a combination of lifestyle factors and the presence of musculoskeletal pain. This could strengthen current evidence about the importance of adhering to a healthy lifestyle and improve understanding of its association with musculoskeletal pain. These findings could help clinicians manage these musculoskeletal pains, by considering the role a lifestyle behavior may have on them.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years (adults), males or females, living in Belgium
* To understand French and/or Dutch
* To be able to provide informed consent
* To have access to the Internet

Exclusion Criteria:

* Age under 18 years
* Inability to complete the questionnaire
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any adult (> 18 years old), male or female, living in Belgium, can complete the questionnaire.
  The study population will include only adults, men and women, living in Belgium, who have access to the Internet.
Sampling Method: Non-Probability Sample
Enrollment: 1188 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Neck pain (in the last 30 days) | Baseline (at the time of completing the questionnaire)
  The presence of neck pain in the last 30 days will be determined using closed questions on pain location, pain intensity, pain-related disability, pain etiology, and pain duration.
Low back pain (in the last 30 days) | Baseline (at the time of completing the questionnaire)
  The presence of low back pain in the last 30 days will be determined using closed questions on pain location, pain intensity, pain-related disability, pain etiology, and pain duration.
Temporomandibular pain (in the last 30 days) | Baseline (at the time of completing the questionnaire)
  The presence of temporomandibular pain in the last 30 days will be determined using the "Temporo-Mandibular Disorders Pain Screener DC-TMD" questionnaire (which consists of 3 questions designed to screen for the presence of temporomandibular pain in the last 30 days) and closed questions on pain-related disability.
Multisite pain (in the last 30 days) | Baseline (at the time of completing the questionnaire)
  The presence of multisite pain in the last 30 days will be determined by the presence of more than one musculoskeletal pain in the last 30 days.
Tobacco consumption | Baseline (at the time of completing the questionnaire)
  Tobacco consumption will be assessed through closed questions about the past and current smoking use, but also about passive smoking. Participants will be separated into 5 groups : daily smokers, occasional smokers, ex-smokers, passive smokers, and non smokers. Only non smokers and non passive smokers will be considered "healthy".
Sleep quality | Baseline (at the time of completing the questionnaire)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-report questionnaire that consists of 19 items related to sleep habits within the past month and 7 clinically relevant domains of sleep difficulties: subjective sleep quality; sleep latency; sleep duration; sleep efficiency; sleep disturbances; use of sleep medication; and daytime dysfunction. Its score ranges from 0 to 21, and a total score > 5 is used to indicate poor sleepers. Participants with a score less than or equal to 5 will be considered "healthy".
Physical activity | Baseline (at the time of completing the questionnaire)
  Physical activity will be assessed using the European Health Interview Survey - Physical Activity Questionnaire (EHIS-PAQ). The EHIS-PAQ is a self-report questionnaire that aims to evaluate how far the population is physically active and assesses PA during work, transportation, leisure time, sports, health-enhancing, and muscle-strengthening activities over a typical week. Participants will be considered "healthy" if they perform leisure-time or sports physical activity at least 150 minutes at moderate intensity or 75 minutes at high intensity per week (or a combination of these intensities), and strength training of the major muscles groups at least 2 days per week.
Consumption of fruits and vegetables | Baseline (at the time of completing the questionnaire)
  Daily consumption of fruits and vegetables will be assessed by asking participants the amount of servings of fruits and vegetables they eat daily. Participants will be considered "healthy" if they consume 5 or more servings of fruits and vegetables per day (e.g., at least 500g/day).
Perceived stress | Baseline (at the time of completing the questionnaire)
  Perceived stress will be assessed using the "Perceived Stress Scale - 10 items" (PSS-10). PSS-10 assesses the imbalance between the individual's perception of the constraints of his environment and his perception of his own ability to cope with them. PSS-10 is a self-report questionnaire of 10 items, in which people are asked to rate on a 5-point scale the extent to which they experienced each of the listed feelings and thoughts, in the past month (from "never" to "very often"). Participants with a total PSS-10 score between 0 and 13 ("low stress") will be considered "healthy".
Body mass index | Baseline (at the time of completing the questionnaire)
  Body Mass Index (BMI) will be assessed by asking participants about their height and weight. Height and weight will be combined to calculate the BMI : weight/height² (kg/m²). Participants with a BMI between 18.5 kg/m² and less than 25 kg/m² will be considered "healthy" (normal weight).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pitance, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No